CLINICAL TRIAL: NCT04146480
Title: The Potential Role of 18F-NaF PET/CT in Diagnosing Cardiac Amyloidosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-17-ES-0807-CTIL
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac amyloidosis patients (Experimental)
  Interventions: Diagnostic Test: F18-NaF PET/CT

INTERVENTIONS:
Diagnostic Test: F18-NaF PET/CT — The scan will be performed on the Discovery 690 Nuclear Medicine Camera. On the day of the scan, the patient will be admitted to the Office of Nuclear Medicine and will be admitted to administrative. Prior to the scan, the subject will undergo a brief interview by a physician or nurse and a 22 G Prefill will be installed on him, through which a 5 millikiric (mCi) of 18 F-NaF will be injected.
  4. An hour after the injection, the PET / CT scan, which will last about 10 minutes, during, the patient is required to lie down and breathe normally.
  5. Upon completion of the scan, will be released without any restrictions.

SUMMARY:
Cardiac amyloidosis is a common cause of refractory cardiomyopathy and heart failure in an adult population. There are several types of cardiac amyloidosis, but two are the most common (1):

A. AL - Light chain sunset.

B. ATTR - Sunset of transthyretin protein. This amyloidosis has two subtypes:

1. Hereditary / familial - due to genetic mutation
2. Senile / Wild-type (WT) - Acquired with age

The main goal of this study is to evaluate cardiac amyloidosis imaging efficiency using 18F-NaF PET / CT and quantification of absorption [in standard uptake value SUVs]. and to compare cardiac amyloidosis imaging using 18F-NaF PET / CT and gamma camera imaging with 99mTc-PYP.

DETAILED DESCRIPTION:
PET imaging has advantages over gamma imaging, including better resolution, faster and easier testing, and the ability to quantify the absorption intensity. These PET capabilities, potentially, detect subtle differences in disease burden between different heart segments and, subsequently, track response to treatment.

Research Duration:

The entire duration of the study will take about one year (or until all participants in the study complete the tests), As part of the study, tests will be conducted for 20 subjects.

Program details and research steps:

* The study is a prospective study.
* The research was done in collaboration with Prof. Eyal Masheni, Director of the Cyclotron and Radiochemistry Unit at Hadassah Hospital, which will provide twenty doses of 18F-NaF.
* For the Cyclotron and Radiochemistry Unit in Hadassah Hospital, a license to operate as a radiopharmaceutical pharmacy on behalf of the Ministry of Health, and thus valid, a blanket approval by the Ministry of Health to use the materials manufactured therein.

Research phases:

1. Patients will undergo clinical and laboratory evaluation, as well as imaging tests, at the discretion of the treating cardiologist, even before being referred for examination within the study. At this stage, patients will be recruited for the study and given an explanation of the tests that will be passed. If necessary, patients will be referred to the Institute of Nuclear Medicine for more information.
2. The test will be performed on the Discovery 690 Nuclear Medicine Camera.
3. On the day of the examination, the examiner will be admitted to the Office of the Institute of Nuclear Medicine and will be admitted to administrative. Prior to the test, the subject will undergo a brief interview by a physician or nurse and a 22 G Prefill will be installed on him, through which a 5 millikiric (mCi) of 18 F-NaF will be injected.
4. An hour after the injection, the PET / CT test, which will last for about 10 minutes, will be performed during which the patient is required to rest comfortably and breathe normally.
5. Upon completion of the mapped examination, the home will be released without any restrictions.
6. Continued clinical follow-up will be done by the attending cardiologist.

ELIGIBILITY:
Inclusion Criteria:

A. Patients undergoing "cardiac amyloidosis clinic" at Tel Aviv Medical Center and there is a clinical suspicion of having cardiac amyloidosis.

B. Patients who performed 99mTc-PYP mapping and signed an informed consent form to perform another imaging test, namely, 18F-NaF PET / CT.

Exclusion Criteria:

None

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2020-07-24 (Estimated)

PRIMARY OUTCOMES:
Evaluating cardiac amyloidosis imaging efficiency using 18F-NaF PET / CT and quantifying the extent of absorption in SUV standard uptake value | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky medial center, Tel Aviv, Israel, Tel Aviv, Central District, Israel

IPD SHARING:
Plan to Share IPD: Undecided